CLINICAL TRIAL: NCT00493753
Title: Feasibility and Safety of Acupuncture for Systemic Lupus Erythematosus
Brief Title: Feasibility and Safety of Acupuncture for Systemic Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: CRCD-ACU-SLE
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The aim of this pilot study was to evaluate whether acupuncture is safe and acceptable to people with systemic lupus erythematosus (SLE). Twenty-four SLE patients were assigned randomly to receive either 10 sessions of acupuncture, 10 sessions of a minimal-needling control intervention, or their usual medical care alone. It was hypothesized that acupuncture would be safe for people with SLE, and that participants would be able to complete their assigned treatment within 5 to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with SLE, 18 years old or older, pain duration at least 3 times per week for at least 3 months, medications and doses stable for the past month, able to speak, read, and understand English, and provide informed consent.

Exclusion Criteria:

* known pregnancy, active uncontrolled organ involvement, steroid dose greater than 10 mg per day, platelets < 100,000, previous course of acupuncture treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-11; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Safety (side effect and adverse event rates), protocol adherence (expected 80% of sessions completed on time) | 6 weeks

SECONDARY OUTCOMES:
pre-post treatment effect size estimates for self-reported pain and fatigue | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Greco, Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC General Clinical Research Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside Center for Integrative Medicine, Pittsburgh, Pennsylvania